CLINICAL TRIAL: NCT06308575
Title: A Phase II Study of Rivoceranib for Patients With Recurrent or Metastatic Olfactory Neuroblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Request--No Patient Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Elevar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0771; NCI-2024-02155 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Olfactory Neuroblastoma; Recurrent Olfactory Neuroblastoma
MeSH Terms: conditions — Esthesioneuroblastoma, Olfactory | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rivoceranib (Experimental): Particpants will take rivoceranib by mouth 1 time each day while on study.
  Interventions: Drug: Rivoceranib

INTERVENTIONS:
Drug: Rivoceranib — Given by PO

SUMMARY:
To learn if rivoceranib can help to control olfactory neuroblastoma. The safety of this drug in participants with olfactory neuroblastoma will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

- To assess the efficacy of rivoceranib in patients with R/M ONB

Secondary Objective:

* To estimate the median duration of response (DOR)
* Time to response
* To estimate the median progression-free survival (PFS)
* To estimate the median overall survival (OS)
* To assess safety of rivoceranib

Tertiary Objective:

- To explore biomarkers that may predict response to therapy

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 years with histology-proven R/M ONB.
2. Not amenable to curative intent surgery or radiotherapy
3. Measurable disease per RECIST 1.1
4. Performance status ECOG of 0 or 1
5. VEGFR-inhibitor naïve (R/M ONB never treated with VEGFR inhibitors)
6. Laboratory measurements, blood counts:

   a) Hemoglobin ≥ 9 g/dL. Red blood cell transfusions are permitted to meet the hemoglobin inclusion criteria b) Absolute neutrophil count ≥ 1 x 109
   * mL c) Platelets ≥ 80 x 109
   * mL
7. Laboratory measurements, renal function:

   a) Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation
8. Laboratory measurements, hepatic function:

   1. AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN in subjects with liver metastases
   2. Total bilirubin ≤ 1.5 x ULN or ≤ 3.0 x ULN and primarily unconjugated if subject has a documented history of Gilbert's syndrome or genetic equivalent
9. Female participants with reproductive potential must practice two effective contraceptive measures for the duration of study drug therapy and for at least 90 days after completion of study therapy. The two birth control methods can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom, copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).
10. Male participants who are sexually active with women with reproductive potential must agree to use contraception for the duration of treatment and for at least 90 days after completion of study therapy.

Exclusion Criteria:

1. Prior radiation therapy (or other nonsystemic therapy) within 2 weeks prior to enrollment
2. Active CNS disease (participants with asymptomatic and stable, treated CNS lesions who have been off corticosteroids, radiation, or other CNS-directed therapy for at least 4 weeks are not considered active)
3. Red blood cell transfusion dependence, defined as requiring more than 2 units of packed red blood cell transfusions during the 4-week period prior to screening. Red blood cell transfusions are permitted during the screening period and prior to enrollment to meet the hemoglobin inclusion criterion.
4. Prior anticancer therapy including, but not limited to, chemotherapy, immunotherapy, or investigational agents within 4 weeks or 5 half-lives prior to rivoceranib treatment
5. Current participation in another interventional clinical study
6. History of previous malignancy other than malignancy treated with curative intent within less than 5 years. Participants with the following diagnoses represents an exception and may enroll if ≥ 1 year with no evidence of active disease before the first dose of the study drug.:

   1. Non-melanoma skin cancers with no current evidence of disease
   2. Melanoma in situ with no current evidence of disease
   3. Localized cancer of the prostate with prostate-specific antigen of <1 ng/mL
   4. Treated or localized well-differentiated thyroid cancer
   5. Treated cervical carcinoma in situ
   6. Treated ductal/lobular carcinoma in situ of the breast
7. Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti-fungal therapy ≤ 10 days prior to administration of investigational product. Participants with known hepatitis B, hepatitis C (HCV), or HIV infection could go on study provided the viral load is undetectable at screening.
8. Participants with poor-controlled arterial hypertension (systolic blood pressure > 140 mmHg and diastolic blood pressure > 90 mmHg) despite standard medical management
9. Participants with Grade II or greater myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (QTc interval ≥ 450 ms in males and ≥ 470 ms in females);
10. Participants with NYHA (see Appendix 5) Class III-IV cardiac insufficiency or LVEF (left ventricular ejection fraction) < 50% by echocardiography;
11. Presence of multiple factors affecting oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction, which significantly affect drug administration and absorption);
12. Urine protein ≥ ++ or 24 h urine protein > 1.0 g as indicated by urinalysis
13. Female subjects who are pregnant or breast-feeding
14. Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Luana Guimaraes De Sousa, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org